CLINICAL TRIAL: NCT05533658
Title: The Effects of VisionPure™ on Indices of Vision Health and Cognitive Function: A Randomized, Double-Blind, Placebo-Controlled, Parallel Pilot Trial.
Brief Title: The Effects of VisionPure™ on Indices of Vision Health and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Collaborators: True Eye Experts - New Tampa (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1221
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2022-10

CONDITIONS: Eye Health; Vision; Cognitive Function
Keywords: Fish Oil; Vitamin D; Antioxidant; Eye Health; Cognitive Function; Vision Health

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VisionPure Dietary Supplement (Experimental): One dose (2 softgel capsules) will be consumed once daily for 60 days. A single dose contains: 976mg fish oil (120mg eicosapentaenoic acid, 610 mg docosahexaenoic acid), 20mg lutein, 4mg zeaxanthin isomers, 25mcg vitamin D3.
  Interventions: Dietary Supplement: VisionPure Dietary Supplement
- Placebo (Placebo Comparator): One dose (2 softgel capsules) will be consumed once daily for 60 days. A single dose contains: 727mg organic sunflower oil, 15mg organic lemon essential oil, 1.5mg vitamin E T-70, 0.7mg natural fish flavor.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: VisionPure Dietary Supplement — Subjects will consume two softgels capsules of the Treatment (VisionPure) once daily for 60 days. At Day 0, they will come in for a Comprehensive Eye Exam, a National Eye Institute Visual Functioning Questionnaire, and a series of Cognitive Function Exams. After 60 days, subjects will return and repeat the same questionnaires and exams from Day 0.
  Arms: VisionPure Dietary Supplement
Dietary Supplement: Placebo — Subjects will orally consume two softgel capsules of Placebo once daily for 60 days. At Day 0, they will come in for a Comprehensive Eye Exam, a National Eye Institute Visual Functioning Questionnaire, and a series of Cognitive Function Exams. After 60 days, subjects will return and repeat the same questionnaires and exams from Day 0.
  Arms: Placebo

SUMMARY:
VisionPure™ is a softgel dietary supplement containing fish oil, lutein, zeaxanthin, and vitamin D. The intent of the VisionPure product is to assist in maintaining eye and cognitive health while helping to provide protection against blue throughout the day. In this pilot trial, approximately 16 participants will be recruited and randomly assigned to experimental and placebo conditions. Participants will consume 1 serving (2 softgels) per day of their respective study condition for 60 days. Prior to and following the 60 day supplementation period, participants will undergo a series of optometry and cognitive examinations to quantify eye health and cognitive function outcomes.

DETAILED DESCRIPTION:
The study design is a randomized, double-blind, placebo-controlled, parallel design, pilot trial. In this pilot trial, approximately 16 participants will be recruited and randomly assigned to experimental and placebo conditions. Participants will consume 1 serving (2 softgels) per day of their respective study condition for 60 days. All study-related procedures will be carried out at 2 locations, The Applied Science and Performance Institute, as well as at True Eye Experts. Both locations are in Tampa, FL. All screening for the study and the signing of all IRB documents will be held at the Applied Science and Performance Institute. Optometry eye examination at Day 0 and Day 60 will be conducted under the supervision of a board-certified O.D. at the True Eye Experts location. Computer-based cognitive assessments using a program called CNS Vital Signs will be carried out at Day 0 and Day 60 at the Applied Science and Performance Institute. The following exams will be carried out: Verbal Memory, Visual Memory, Composite Memory, and Cognitive Attention.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18-40 years
* English literate
* Willing to sign informed consent form

Exclusion Criteria:

* Current cataracts or prior cataract extraction
* Glaucoma
* Uveitis
* Macular hole or traction
* Retinitis pigmentosa
* Significant epiretinal membrane
* Dry eye syndrome of any form
* LASIK procedure
* Diagnosed concussion within the last 6 months
* Optic neuropathy
* Neurological disease
* Metabolic disease
* Cardiovascular disease
* Renal disease
* History of previous ocular surgery, trauma, intraocular injections or photocoagulation
* Vitamin D3, omega fatty acids, or fish oil supplementation with the last 6 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Change in Ganglion Cell Complex Thickness | Day 0, Day 60
  Diagnostic Procedure: Retinal Optical Coherence Tomography
Change in Central Retinal Thickness | Day 0, Day 60
  Diagnostic Procedure: Retinal Optical Coherence Tomography
Change in Intraocular Pressure | Day 0, Day 60
  Diagnostic Procedure: Retinal Optical Coherence Tomography

SECONDARY OUTCOMES:
Change in Visual Acuity | Day 0, Day 60
  Determines the clarity of your distance vision according to the Snellen Chart.
Change in Color Vision | Day 0, Day 60
  Determines the normality of or defectiveness of color vision. Reference Range: 1 to 11 according to Ishihara Plates (>10 is normal, 7 or <7 is deficient).
Change in Verbal Memory | Day 0, Day 60
  How well can an individual recognize, remember, and recall words.
Change in Visual Memory | Day 0, Day 60
  How well can in individual recognize, remember, and recall a combination of words and images.
Change in Composite Memory | Day 0, Day 60
  How well an individual can recognize, remember, and recall a combination of words and images.
Change in Cognitive Attention | Day 0, Day 60
  The ability to handle multiple tasks at once and shift attention.

OTHER OUTCOMES:
Changes in National Eye Institute Visual Functioning Questionnaire - 25 (VFQ-25) | Day 0, Day 60
  Subjective/Self-Reported Eye Health Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Wilson, Ph.D., Principal Investigator — The Applied Science and Performance Institute
Locations (3):
- United States (3):
  - True Eye Experts - Lutz, Lutz, Florida
  - Applied Science and Performance Institute, Tampa, Florida
  - True Eye Experts - New Tampa, Tampa, Florida